CLINICAL TRIAL: NCT06050109
Title: A Multicenter, Open-label, Non-randomized Controlled Real World Study Comparing the Benefits of Continued Use of Ovarian Function Suppression After 5 Years
Brief Title: The Benefits of Continued Use of Ovarian Function Suppression After 5 Years
Status: Recruiting | Type: Observational
Sponsor: Hongmei Zheng, PhD (Other)
Responsible Party: Sponsor-Investigator, Hongmei Zheng, PhD, vice director, Hubei Cancer Hospital
Organization: Hubei Cancer Hospital (Other)
Other Study IDs: HBCHBCC001
Record Dates: First submitted 2023-09-17; First posted 2023-09-22 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer Female; Endocrine Therapy
Keywords: ovarian function suppression; Hormone receptor (HR) positive; HER2 negative; early breast cancer; prolonged therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- OFS continues to use after 5 years: HR-positive premenopausal female patients whose doctors believe that they can benefit from continued use of OFS after 5 years should be included in the trial group.
  Interventions: Drug: OFS continues to use group after 5 years use; Diagnostic Test: Immunohistochemical detection of HR status
- OFS discontinues to use after 5 years: The control group did not need to continue to use OFS, either leuprolide or goserelin

INTERVENTIONS:
Drug: OFS continues to use group after 5 years use — Patients included in the group continued or discontinued to use goserelin or leuprolide after 5 years use.
  Other Names: OFS discontinues to use group after 5 years use
  Groups: OFS continues to use after 5 years
Diagnostic Test: Immunohistochemical detection of HR status — Enrolled patients must be HR-positive premenopausal breast cancer patients
  Groups: OFS continues to use after 5 years

SUMMARY:
To observe and evaluate the clinical efficacy and safety of continuous use of OFS for premenopausal patients with early breast cancer after 5 years use of OFS.

This study is a multicenter, prospective, observational, non randomized controlled, open-label real world study based on hospital medical record system data, aimed at evaluating the benefits of continuing to use OFS after 5 years of use. The retrospective analysis plan includes patient data from September 1, 2023 to September 1, 2026. Join two cohorts: the continued use group and the discontinued use group after 5 years of OFS, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with early primary breast cancer
* Female aged 18-60 years (including 18 year and 60 year)
* Hormone receptor (HR) positive HER2 negative
* Receive 5 years of OFS treatment
* ECOG score 0-1
* Voluntarily join this study and sign the informed consent form;
* The researcher believes that it can benefit.

Exclusion Criteria:

* The patient is receiving treatment that affects OFS at the same time The patient has received OFS treatment for less than 5 years
* Central nervous system metastases with known obvious symptoms, such as headache, cerebral edema, blurred vision
* Invasive metastases with known obvious symptoms
* Invasive metastases with known obvious symptoms
* Doctors think it is not suitable for inclusion

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women who are diagnosed as early breast cancer and have received 5 years treatment of OFS.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
invasive disease-free survival | 5 years
  The main effect evaluation index was invasive disease-free survival (iDFS)

SECONDARY OUTCOMES:
Overall survival | 5 years
  Overall survival for years, which means the rate of patients alive in the whole patients at the same group will be calculated with kaplan meier survival curves.

OTHER OUTCOMES:
Quality of life score | 5 years
  Quality of life score was evaluated by European Organization of Research and treatment of Cancer-Questionnaire of Life Quality-C30 Version 3 (EORTC-QLQ-C30 V3), which conduct a series of questions about the patients' physical condition, activity of daily life, adverse reaction and mood condition. The range in the questionnaire for the score is from 1 to 4, in which 1 stands for having no discomfort and 4 stands for having great discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Hongmei Zheng, Doctor, Principal Investigator — Study Principal Investigator
Locations (1):
- Wu Xinhong, Wuhan, Hubei, China